CLINICAL TRIAL: NCT00658671
Title: An Open-Label, Dose-Escalation, Safety, and Pharmacokinetic Study of ENMD-2076 Administered Orally to Patients With Advanced Cancer
Brief Title: A Dose-Escalation Study of ENMD-2076 Administered Orally to Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2076-CL-001
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — ENMD 2076

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Dose-escalation
  Interventions: Drug: ENMD-2076
- 2 (Experimental): Advanced cancer, excluding patients with colorectal or ovarian cancers
  Interventions: Drug: ENMD-2076
- 3 (Experimental): Recurrent or resistant epithelial ovarian cancer
  Interventions: Drug: ENMD-2076
- 4 (Experimental): Colorectal cancer patients who have progressed and/or failed on irinotecan- and oxaliplatin-based regimens
  Interventions: Drug: ENMD-2076

INTERVENTIONS:
Drug: ENMD-2076 — Capsules, daily dosing in 28 day cycles

SUMMARY:
A dose-escalation trial designed to assess the safety and tolerability of treatment with ENMD-2076 administered orally over a range of doses in patients with advanced cancer that is refractory to current treatment or for which no curative therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Have histologic proof of advanced cancer that has progressed after treatment and has no standard therapy that is curative or provides clinical benefit.
* Meet the modified RECIST Criteria or have disease that can be followed for clinical benefit.
* Are greater than or equal to 18 years of age.
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Total bilirubin ≤ ULN
* Creatinine ≤ 1.5 x ULN
* Absolute neutrophil count ≥ 1500 cells/mm3
* Platelets ≥ 100,000/mm3
* Hemoglobin ≥ 9.0 g/dL
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Agree to use effective contraceptive methods prior to study entry, during study participation, and for at least 30 days after the last administration of study medication.
* Have the ability to understand the requirements of the study, provide written informed consent which includes authorization for release of protected health information, abide by the study restrictions, and agree to return for the required assessments.

Exclusion Criteria:

* Women who are pregnant or nursing.
* Have received radiotherapy or chemotherapy less than two weeks prior to first dose of study medication and have not recovered from all acute toxicities from prior treatments.
* Have participated in any clinical trial involving conventional or investigational drugs within 28 days prior to initiation of ENMD-2076 dosing.
* Have active, acute, or chronic clinically significant infections.
* Have uncontrolled severe hypertension or congestive heart failure.
* Have active angina pectoris or recent myocardial infarction (within 6 months).
* Have chronic atrial fibrillation or QTc of greater than 470 msec.
* Have had major surgery within 21 days of starting therapy.
* Have planned surgical treatment of tumor(s)
* Have additional uncontrolled serious medical or psychiatric illness.
* Have any medical condition that would impair the administration of oral agents including significant bowel resection, inflammatory bowel disease or uncontrolled nausea or vomiting.
* Have a 2+ protein by urinalysis or a history of nephrotic syndrome.
* Known central nervous system metastasis.
* Have history of deep vein thrombosis or pulmonary embolus, unless they are receiving therapeutic anticoagulation with warfarin or low-molecular-weight heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ENMD-2076 | Throughout study treatment

SECONDARY OUTCOMES:
Plasma PK | Throughout study treatment
Evidence of benefit (tumor response, clinical benefit, or tumor marker improvement, if appropriate) | Throughout study treatment

CONTACTS AND LOCATIONS:
Overall Officials: William Gannon, MD, MBA, Study Director — CASI Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Dana Farber/Harvard Cancer Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Diamond JR, Bastos BR, Hansen RJ, Gustafson DL, Eckhardt SG, Kwak EL, Pandya SS, Fletcher GC, Pitts TM, Kulikowski GN, Morrow M, Arnott J, Bray MR, Sidor C, Messersmith W, Shapiro GI. Phase I safety, pharmacokinetic, and pharmacodynamic study of ENMD-2076, a novel angiogenic and Aurora kinase inhibitor, in patients with advanced solid tumors. Clin Cancer Res. 2011 Feb 15;17(4):849-60. doi: 10.1158/1078-0432.CCR-10-2144. Epub 2010 Dec 3. PMID 21131552